CLINICAL TRIAL: NCT05012098
Title: Phase 2 Study of Bintrafusp Alfa in Recurrent/Metastatic Olfactory Neuroblastoma (BARON).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charalampos Floudas, MD, DMSc, MS, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000030; 000030-C
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Olfactory Neuroblastoma; Esthesioneuroblastoma; Neoplasm of the Nasal Cavity
Keywords: ONB; M7824; nasal tumor
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory; Nose Neoplasms | interventions — Ibuprofen; Positron-Emission Tomography; Tomography, X-Ray Computed; Radionuclide Imaging; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1: Treatment with Bintrafusp Alfa (Experimental): Treatment with Bintrafusp alfa
  Interventions: Drug: Bintrafusp alfa/M7824; Drug: Ibuprofen; Diagnostic Test: PET scan; Diagnostic Test: CT scan; Procedure: Tumor tissue biopsy; Diagnostic Test: Brain MRI; Diagnostic Test: Dotate scan; Diagnostic Test: PET FDG scan; Diagnostic Test: Nuclear bone scan; Diagnostic Test: EKG

INTERVENTIONS:
Drug: Bintrafusp alfa/M7824 — Participants will be treated with bintrafusp alfa 1200 mg every 2 weeks for 26 doses.
  Other Names: M7824
Drug: Ibuprofen — 400 mg or comparable non-steroidal anti-inflammatory drugs (NSAIDs) dose up to 2 hours before and 8 hours after the start of each dose for prophylaxis of flu-like symptoms.
  Other Names: Advil; Advil Migraine
Diagnostic Test: PET scan — Screening
  Other Names: Positron emission tomography scan
Diagnostic Test: CT scan — Screening
  Other Names: Computed tomography scan
Procedure: Tumor tissue biopsy — Baseline, and subsequent weeks as stipulated in the study calendar.
  Other Names: Tumor tissue bx
Diagnostic Test: Brain MRI — Baseline
  Other Names: Brain magnetic resonance imaging
Diagnostic Test: Dotate scan — Baseline
  Other Names: Ga-68 dotatate positron emission tomography/computed tomography scan
Diagnostic Test: PET FDG scan — Baseline
  Other Names: fludeoxyglucose-18 (FDG) positron emission tomography (PET) scan
Diagnostic Test: Nuclear bone scan — Baseline
Diagnostic Test: EKG — Baseline
  Other Names: Electrocardiogram

SUMMARY:
Background:

Olfactory neuroblastoma (ONB) is a rare cancer of the nasal cavity. At diagnosis, it is usually locally advanced. It tends to spread to the neck. Sometimes it spreads to the lungs and bones. Researchers want to find a better way to treat it.

Objective:

To learn if giving immunotherapy drug bintrafusp alfa can help ONB shrink or disappear.

Eligibility:

People aged 18 years and older diagnosed with recurrent or metastatic ONB that has not responded to standard treatment.

Design:

Participants will be screened with a medical history, blood and urine tests, and physical exam. Their ability to perform their normal activities will be assessed. They will have an electrocardiogram to evaluate their heart. They will have imaging scans and/or a nuclear bone scan, as needed. For some scans, they may receive a contrast dye.

Some screening tests will be repeated during the study.

Participants will receive bintrafusp alfa once every 2 weeks for 26 doses. They will get it intravenously over 60 minutes. They may get other medicines to prevent side effects. They will complete health questionnaires. Visits will last 4-6 hours.

Participants may have optional tumor biopsies.

Participants will have an end of treatment visit within 7 days after they stop taking the study drug. About 28 days after treatment ends, they will have a safety visit. They will have follow-up visits every 3 months for the first year, then every 6 months for years 2-5, and then once a year after that for the rest of their life. If their disease progresses, they may be eligible for re-treatment with the study drug

DETAILED DESCRIPTION:
Background:

Olfactory neuroblastoma (ONB, also known as esthesioneuroblastoma), is a rare malignant neoplasm of the nasal cavity. At diagnosis, ONB is often locally advanced. It tends to invade locally and has high rates of regional spread to the neck, and distally to the lungs and bones. The 10-year survival rate for ONB is reported at 46%.

Standard of care treatment is surgical resection followed by adjuvant radiation. In advanced unresectable or metastatic cases, systemic chemotherapy is used off label, with agent selection based on published case series. Genomic profiling of ONB has not yet informed the utilization of an appropriate molecularly targeted treatment.

High programmed death-ligand 1 (PD-L1) expression by immunohistochemistry was shown in ONB tumor samples, providing a rationale for immune checkpoint blockade in ONB. In addition, high expression of transforming growth factor beta (TGF-beta) ligands has been identified in ONB, implying that additional benefit may be achieved by combination of checkpoint blockade with TGF-beta inhibition.

Bintrafusp alfa is a novel bifunctional fusion protein composed of a blocking monoclonal antibody against PD-L1 fused with the soluble extracellular domain of the human TGF-beta receptor II (TGF-betaRII), acting as a decoy target for TGF-beta. The safety profile of bintrafusp alfa in clinical trials to date has been shown to be manageable.

Objective:

To assess the objective response rate (ORR) to bintrafusp alfa in participants with recurrent/metastatic ONB, immune checkpoint-naive (CN)

Eligibility:

Participants must have histologically confirmed recurrent or metastatic ONB, not amenable to potentially curative local therapies.

Participants should have received at least one line of systemic therapy including a platinum agent, with evidence of disease progression clinically or radiographically.

Presence of >= 1 lesion measurable by Response Evaluation Criteria in Solid Tumors, (RECIST) 1.1 criteria

Age >= 18 years, men and women

Adequate organ function, and without serious comorbidity (e.g., autoimmune disease), that would preclude concurrent systemic treatment.

Design:

Single-institution, single-arm Phase II trial to determine overall response rate (ORR) in participants with recurrent/metastatic ONB treated with bintrafusp alfa.

Participants will be treated with bintrafusp alfa 1200 mg every 2 weeks for 26 doses.

The trial will initially enroll 12 checkpoint-naive (CN) participants; if responses are observed in one or more participants, the second stage will enroll another 9 CN participants to define the response rate to bintrafusp alfa, for a total of 21 CN participants.

An additional cohort of checkpoint-resistant (CR) participants will be enrolled and evaluated separately. Initially 5 CR participants will be enrolled; if responses are observed in one or more participants, the second stage will enroll another 3 participants, for a total of up to 8 CR participants. Accrual for CR participants will end when the preset number of CN participants has been accrued.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histologically or cytologically confirmed recurrent or metastatic olfactory neuroblastoma (ONB) not amenable to potentially curative local therapies. Review of tissue samples by Pathology at the National Institutes of Health (NIH) is preferred.
2. Participants must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. A previously treated lesion by radiotherapy can be chosen as the target lesion only if progression in the respective lesion has been demonstrated during or following radiotherapy.
3. Participants should have received at least one line of systemic therapy including a platinum agent, with evidence of disease progression clinically or radiographically.
4. Men or Women >=18 years of age on day of signing informed consent. Because no dosing or adverse event data are currently available on the use of bintrafusp alfa in participants <18 years of age, children are excluded from this study.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) =<2.
6. Participants must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) >=1,500/mcL
   * Hemoglobin >=9 g/dL (transfusions allowed)
   * Platelets >=100,000/mcL
   * Serum Creatinine <= 1.5 x upper limit of normal (ULN) OR Measured creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula may be used to estimate CrCl/eGFR >=30 mL/min/1.73m^2 for participant with creatinine levels > 1.5 x institutional ULN
   * Serum total bilirubin <=1.5 x upper limit of normal (ULN) OR Direct bilirubin <=ULN for participants with total bilirubin levels >1.5 x ULN
   * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) <=2.5 x ULN
7. The effects of immunotherapy on the developing human fetus are unknown. Therefore, participants must use effective methods of contraception (such as implants, injectables, combined oral contraceptives, intrauterine device (IUDs), sexual abstinence or vasectomized partner).

   * Women of child-bearing potential (WOCBP: any woman who has experienced menarche and has not had hysterectomy or bilateral oophorectomy or is not postmenopausal (amenorrheic 12 months or more following cessation of exogenous hormonal treatments; if <50 years old need follicle stimulating hormone (FSH) in the post-menopausal range)) must agree to use highly effective contraception prior to study entry and for up to 65 days following the last dose of study treatment.
   * Men must agree to use highly effective contraception prior to study entry and up to 125 days following the last dose of study treatment.
   * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
8. Participants with bone metastases or hypercalcemia on intravenous bisphosphonate treatment, zolendronic acid, denosumab, or similar agents are eligible to participate and may continue this treatment.
9. Participants with treated central nervous system (CNS) ONB lesions are eligible if follow-up brain imaging after at least a month following central nervous system (CNS)-directed therapy shows no evidence of progression.
10. Participants with new or progressive non-intraparenchymal CNS ONB lesions are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
11. Human immunodeficiency virus (HIV)-positive participants must have cluster of differentiation 4 (CD4) count >= 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman's disease within 12 months prior to enrollment.
12. For participants with serological evidence of chronic hepatitis B virus (HBV) infection, the HBV deoxyribonucleic acid (DNA) viral load must be undetectable on suppressive therapy, if indicated.
13. For participants with serological evidence of hepatitis C virus (HCV) infection, the HCV ribonucleic acid (RNA) viral load must be negative to be eligible for study participation.
14. Ability of participant to understand and the willingness to sign a written informed consent document.
15. Must co-enroll in the following two studies. A separate inform consent will be obtained from participant for these studies.

    * 21-C-0009: A Natural History Study of Children and Adults with Olfactory Neuroblastoma, and
    * 18-DC-0051: Biospecimen procurement for NIDCD clinical protocols

EXCLUSION CRITERIA:

1. Anticancer treatment, concurrent or prior (chemotherapy, monoclonal antibody, cytokine therapy, immune therapy, targeted small molecule therapy) or any investigational drug, within 4 weeks or 5 half-lives (whichever shorter) prior to the first drug administration. All residual treatment-related toxicities must have resolved or be minimal and not constitute a safety risk. Note: Palliative radiotherapy is permitted concurrently or within the pretreatment period. Subjects receiving bisphosphonates or denosumab are eligible provided treatment was initiated at least 14 days before treatment.
2. Participants who received prior checkpoint blockade therapy and were taken off treatment for serious adverse events related to immuno-therapy are excluded.
3. Major surgery within 4 weeks prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).
4. Active or prior documented autoimmune or inflammatory diseases that might deteriorate on immunostimulatory agent (including colitis or Crohn's disease, systemic lupus erythematosus, sarcoidosis, vasculitis, Grave's disease, hypophysitis, uveitis, rheumatoid arthritis etc.), except the following:

   * Type I diabetes mellitus
   * Chronic skin conditions that do not require systemic therapy (including eczema, vitiligo, alopecia, psoriasis)
   * Hypothyroidism (e.g., post-Hashimoto thyroiditis) stable, on hormone replacement
   * Mild autoimmune disease not active in the last 5 years may be eligible after consultation with the principal investigator.
5. Current use of immunosuppressive medication within 14 days before the first dose of the study medication, except the following:

   * Intranasal, inhaled, topical glucocorticoids; locally injected glucocorticoids (i.e. intra-articular, intra-ocular)
   * Systemic glucocorticoids at physiologic doses (generally <= 10 mg prednisone or equivalent per day)
   * Glucocorticoids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.
6. Uncontrolled intercurrent chronic or acute illness including, but not limited to the following, that may limit interpretation of results or increase risk to the participant in the judgment of the investigator:

   * Bleeding diathesis or recent (<3 months) clinically significant bleeding event.
   * Prior organ transplantation including allogenic stem-cell transplantation
   * Impaired cardiovascular function or clinically significant cardiovascular disease, including, but not limited to, any of the following:

     * cerebral vascular accident/stroke (< 3 months prior to enrollment),
     * acute coronary syndromes (including myocardial infarction < 6 months prior to enrollment, unstable angina),
     * Congestive Heart Failure (>= New York Heart Association Classification Class III); CHF Class II must have been stable for 3 months prior to enrollment
     * history or presence of clinically significant cardiac arrhythmia including resting bradycardia, uncontrolled atrial fibrillation or paroxysmal supraventricular tachycardia (controlled arrhythmias, e.g., stable atrial fibrillation, may be allowed at the discretion of the investigator),
     * history of myocarditis
   * History of idiopathic pulmonary fibrosis, drug-induced or idiopathic pneumonitis, active interstitial lung disease, blood oxygen saturation <90% at rest (on ambient air).
   * Clinically significant hepatic disease.
   * Active infection requiring systemic therapy (minor infections may be allowed at the discretion of the investigator).
7. Subjects unwilling to accept blood products as medically indicated.
8. Vaccination with live vaccines within 4 weeks of the first dose of treatment and while on study is prohibited. Inactivated vaccines may be administered.
9. History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to bintrafusp alfa. Participants with history of severe hypersensitivity reaction to monoclonal antibodies (grade >= 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5) will be evaluated by the allergy/immunology team prior to enrollment.
10. History of second malignancy within 3 years of enrollment except for the following: adequately treated localized basal cell or squamous skin cancer, cervical carcinoma in situ, superficial bladder cancer, other localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk chronic lymphocytic leukemia (CLL).
11. Pregnant or breastfeeding women are excluded from this study because the study medications have not been tested in pregnant women and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study medications, breastfeeding should be discontinued if the mother is treated on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Haque F, Carrasquillo JA, Turkbey EB, Mena E, Lindenberg L, Eclarinal PC, Nilubol N, Choyke PL, Floudas CS, Lin FI, Turkbey B, Harmon SA. An automated pheochromocytoma and paraganglioma lesion segmentation AI-model at whole-body 68Ga- DOTATATE PET/CT. EJNMMI Res. 2024 Nov 5;14(1):103. doi: 10.1186/s13550-024-01168-5. PMID 39500789
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000030-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1/Arm 1: Treatment With Bintrafusp Alfa -Immune Checkpoint; Cohort 2/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint Blockade Resistant (ICB-R): Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
Period: Overall Study
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa -Immune Checkpoint | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint Blockade Resistant (ICB-R)
Started | 9 | 2
Completed Study | 1 | 0
Lost to Further Follow-up | 1 | 0
Completed | 1 | 0
Not Completed | 8 | 2
Not completed — Disease progression | 5 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discontinuation per protocol | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1/Arm 1: Treatment With Bintrafusp Alfa-Immune Checkpoint; Cohort 2/Arm 1: Treatment With Bintrafusp Alfa- Immune Checkpoint Blockade Resistant (ICB-R): Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
- Total: Total of all reporting groups
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa-Immune Checkpoint | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa- Immune Checkpoint Blockade Resistant (ICB-R) | Total
Number analyzed (Participants) | 9 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 9
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.11 (7.57) | 53 (2.83) | 58 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: ORR is defined as the percentage of evaluable participants who experience a response evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 reported along with a 95% two-sided confidence interval. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Cycle 1 (28 days)
Population: Only the immune checkpoint-naïve participants will be included in the primary endpoint analysis as pre-specified by the protocol. 8/9 participants were analyzed because one participant was non-evaluable for response
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint: Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint
Number analyzed (Participants) | 8
Percentage of participants
  Complete Response | 0 [0 to 0]
  Partial Response | 0 [0 to 0]
  Stable Disease | 37.5 [8.5 to 75.5]
  Progressive Disease | 62.5 [24.5 to 91.5]

2. Secondary Outcome: Number of Participants Who Experience a Toxicity Related to Bintrafusp Alfa (M7824), by Grades (1, 2, 3, 4 and/or 5) and Type of Toxicity
Description: The number of participants who experience toxicity, by grade and type of toxicity related to Bintrafusp alfa (M7824) was assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Participants in Cohort 1/Arm 1 With Grade 1 Toxicity; Participants in Cohort 1/Arm 1 With Grade 2 Toxicity; Participants in Cohort 1/Arm 1 With Grade 3 Toxicity; Participants in Cohort 1/Arm 1 With Grade 4 Toxicity; Participants in Cohort 1/Arm 1 With Grade 5 Toxicity: Cohort 1/Arm 1: Treatment with Bintrafusp Alfa:
  Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
- Participants in Cohort 2/Arm 1 With Grade 1 Toxicity; Participants in Cohort 2/Arm 1 With Grade 2 Toxicity; Participants in Cohort 2/Arm 1 With Grade 3 Toxicity; Participants in Cohort 2/Arm 1 With Grade 4 Toxicity; Participants in Cohort 2/Arm 1 With Grade 5 Toxicity: Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
Arm/Group | Participants in Cohort 1/Arm 1 With Grade 1 Toxicity | Participants in Cohort 1/Arm 1 With Grade 2 Toxicity | Participants in Cohort 1/Arm 1 With Grade 3 Toxicity | Participants in Cohort 1/Arm 1 With Grade 4 Toxicity | Participants in Cohort 1/Arm 1 With Grade 5 Toxicity | Participants in Cohort 2/Arm 1 With Grade 1 Toxicity | Participants in Cohort 2/Arm 1 With Grade 2 Toxicity | Participants in Cohort 2/Arm 1 With Grade 3 Toxicity | Participants in Cohort 2/Arm 1 With Grade 4 Toxicity | Participants in Cohort 2/Arm 1 With Grade 5 Toxicity
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 2 | 2 | 2 | 2 | 2
Participants
  Serious: Metabolism and nutrition disorders: Immune-mediated diabetes | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Esophageal hemorrhage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Acute kidney injury | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Anemia | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Non-serious: Arthralgia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Aspartate aminotransferase increased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Atrioventricular block first degree | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Bruising | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Cardiac troponin I increased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Constipation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Diarrhea | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Non-serious: Dry eye | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Electrocardiogram T wave abnormal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Epistaxis | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Non-serious: Flu like symptoms | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Folliculitis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Headache | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Hemorrhoidal hemorrhage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Hyperhidrosis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Hypothyroidism | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Insomnia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Lipase increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Non-serious: Neoplasms benign, malignant and unspecified: Keratoacanthoma | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Non-serious: Oral dysesthesia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Oral hemorrhage | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Non-serious: Pharyngeal mucositis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Platelet count decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Pneumonitis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Pruritus | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Non-serious: Rash maculo-papular | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-serious: Skin hypopigmentation: Vitiligo | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first treatment to the date of death (any cause) using the Kaplan-Meier method.
Time Frame: Through study completion, an average of 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa-Immune Checkpoint | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa- Immune Checkpoint Blockade Resistant (ICB-R)
Number analyzed (Participants) | 9 | 2
Months | NA [7.9 to NA] — The median and upper confidence interval are not estimable because there are not enough events within the follow-up period. | 2.1 [2.1 to NA] — The upper confidence interval is not estimable because there are not enough events within the follow-up period.

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time measurement for complete response (CR) or partial response (PR) (whichever is first recorded) until the first documented date of progressive disease (PD) or death. ORR was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 using the Kaplan-Meier method and reported along with a 95% two-sided confidence interval. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions.
Time Frame: Through treatment completion, an average of 1 year
Population: No participants experienced Complete or Partial Response therefore Duration of Response could not be assessed.
Groups:
- Cohort 2/Arm 1: Treatment With Bintrafusp Alfa-Immune Checkpoint Blockade Resistant (ICB-R): Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa-Immune Checkpoint | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa-Immune Checkpoint Blockade Resistant (ICB-R)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first, using the Kaplan-Meier method and reported along with a 95% confidence interval. Disease progression was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is at least a 20% increase in the sum of the diameters of target lesions.
Time Frame: Through treatment completion, an average of 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint Blockade Resistant (ICB-R)
Number analyzed (Participants) | 9 | 2
Months | 9.3 [1.8 to NA] — The upper confidence interval is not estimable due to the limited number of progression events. | 2.99 [0.9 to NA] — The upper confidence interval is not estimable due to the limited number of progression events.

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events were monitored/assessed from first drug administration through 30 days after the last dose of study drug is administered, an average of 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa - Immune Checkpoint Blockade Resistant (ICB-R)
Number analyzed (Participants) | 9 | 2
Participants | 9 | 2

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed an average of 6 months. Adverse Events were monitored/assessed from first drug administration through 30 days after the last dose of study drug is administered, an average of 6 months.
Groups:
- Cohort 1/Arm 1: Treatment With Bintrafusp Alfa; Cohort 2/Arm 1: Treatment With Bintrafusp Alfa: Treatment with Bintrafusp alfa
  Bintrafusp alfa/M7824: Participants will be treated with bintrafusp alfa 1200 mg intravenous over 60 minutes (+/- 20 minutes) once every 2 weeks for 26 doses.
Arm/Group | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/2
Other Adverse Events (participants affected / at risk) | 9/9 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa (N=9) | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa (N=2)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Corneal perforation (Eye disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, Immune-mediated diabetes (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Arm 1: Treatment With Bintrafusp Alfa (N=9) | Cohort 2/Arm 1: Treatment With Bintrafusp Alfa (N=2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (6) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 2 (3) | 0 (0)
Gastrointestinal disorders - Other, specify - Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (2)
Localized edema (General disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify - Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (8) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify - Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify - (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Milia cysts; Basal skin carcinoma
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1)
Eye disorders - Other, specify - Corneal perforation (Eye disorders) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify - Immune-mediated diabetes (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 1 (1) — Keratoacanthoma: 5; Basal skin cancer: 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT05012098/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT05012098/ICF_001.pdf